CLINICAL TRIAL: NCT03753152
Title: A Multicenter Randomized, Evaluator-Blinded, Active Controlled Design Study to Evaluate the Safety and Effectiveness of Neuramis® Deep Lidocaine Compared to YVOIRE® Volume Plus for Correction of Nasolabial Folds
Brief Title: Neuramis® Deep Lidocaine Compared to YVOIRE® Volume Plus for Correction of Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT07-CN16NLF701
Record Dates: First submitted 2018-11-22; First posted 2018-11-26 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational medical device (Experimental): Neuramis® Deep Lidocaine
  Interventions: Device: experimental
- Comparator device (Active Comparator): YVOIRE® Volume Plus
  Interventions: Device: comparator

INTERVENTIONS:
Device: experimental — Neuramis® Deep Lidocaine
  Arms: Investigational medical device
Device: comparator — YVOIRE® Volume Plus
  Arms: Comparator device

SUMMARY:
This clinical investigation is a randomized, evaluator-blind, active controlled, noninferiority study to evaluate the effectiveness and safety of Neuramis® Deep Lidocaine when compared with YVOIRE® Volume Plus.

DETAILED DESCRIPTION:
Males or females between 18 and 75 years of age, who want to correct both NLFs with 3 or 4 points in the WSRS and who provided written informed consent are to be included in the investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 75 years of age.
2. Subjects who desire correction of bilateral NLFs that are rated as 3 or 4 points on the WSRS.

Exclusion Criteria:

1. Subjects who have received anticoagulation, antiplatelet, or thrombolytic medications, anti inflammatory medications.
2. Subjects who had soft tissue augmentation, medium or deep peeling, or dermal photorejuvenation on the lower inferior orbital rim for wrinkle correction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
WSRS improvement rate at Week 24 | Week 24
  WSRS improvement rate at Week 24

SECONDARY OUTCOMES:
Change of WSRS from Week 4, 12, 24, 36, and 52 | Week 4, 12, 24, 36, and 52
  Change of WSRS from Week 4, 12, 24, 36, and 52
WSRS improvement rate on Week 4, 12, 36, and 52 | Week 4, 12, 36, and 52
  WSRS improvement rate on Week 4, 12, 36, and 52
GAIS improvement rate on Week 4, 12, 24, 36, and 52 | Week 4, 12, 24, 36, and 52
  GAIS improvement rate on Week 4, 12, 24, 36, and 52

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua XU, Principal Investigator — Huashan Hospital
Locations (1):
- HuaShan hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No